CLINICAL TRIAL: NCT01640158
Title: BRAVE Trial: Broad-spectrum Cognitive Remediation Available to Veterans: Effects of a Brain Plasticity-based Program in Mild Traumatic Brain Injury (mTBI)
Brief Title: Broad-spectrum Cognitive Remediation: Effects of a Brain Plasticity-based Program in Mild Traumatic Brain Injury
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency); VA Connecticut Healthcare System (U.S. Federal Agency); VA Boston Healthcare System (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPI-1002-11
Record Dates: First submitted 2012-07-10; First posted 2012-07-13 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Brain Injury
Keywords: mild Traumatic Brain Injury; Cognitive remediation; computer
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training, up to 65 hours
  Interventions: Other: Computerized Plasticity-based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training, up to 65 hours
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-based Adaptive Cognitive Training — Computerized plasticity-based adaptive cognitive training, up to 65 hours
  Arms: Experimental Treatment
Other: Commercially available computerized training — Commercially available computerized training, up to 65 hours
  Arms: Active Comparator

SUMMARY:
The primary objective of this study is to evaluate the effects of plasticity-based, adaptive cognitive remediation on the cognitive abilities, functional status and quality of life of soldiers and veterans diagnosed with persistent post-concussive symptoms (PPCS) following a mild traumatic brain injury (mTBI, also referred to as a concussion, or blast exposure), as compared to a computer-based control.

DETAILED DESCRIPTION:
This study is a multi-site, prospective, parallel arm, double-blind, randomized, controlled clinical trial to assess the safety and efficacy of plasticity-based, adaptive, computerized cognitive remediation treatment versus a computer-based control. Both the study and the cognitive remediation treatments meet the criteria of Non-Significant Risk.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 - 50 years of age at the time of consent
2. Subjects must have a diagnosis of mTBI
3. Subjects must have persistent cognitive dysfunction confirmed by an objective measure (as recommended by the ICD-10 definition for post-concussion syndrome) or a subjective measure (as recommended by the DSV-IV definition of post-concussional disorder).
4. Subjects must be at least three months out from their most recent TBI, concussion, and/or blast exposure to minimize the effects of spontaneous recovery, as verified through participant interview.
5. Subjects must be fluent English speakers.
6. Subjects must have adequate sensorimotor capacity to perform the program in the judgment of the consenting clinician.

Exclusion Criteria:

1. Subjects must not have a history of penetrating head wounds or a diagnosis of moderate or severe TBI.
2. Subjects must not be in-patients.
3. Subjects must not have a diagnosis of an illness or condition with known cognitive consequences (e.g., schizophrenia, bipolar disorder, cancer, multiple sclerosis).
4. Subjects must not show suicidal ideation as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS).
5. Subjects must now show signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs) during any in person visit.
6. Subjects must not have clinically significant visual field deficits noted by the consenting staff member by direct observation or by medical history.
7. Subjects must not be judged to be lacking effort.
8. Subjects must not have problems performing assessments or comprehending or following spoken instructions.
9. Subjects must not be enrolled in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device, or behavioral treatment for TBI that could affect the outcome of this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | After three months of training
  Between-group magnitude of change in composite score with the measure constructed from Rey Auditory Verbal Learning Test (RAVLT) sum of trials 1-5 (immediate verbal memory), RAVLT delayed verbal recall, the Ruff Light Trails Test (RULIT) sum of trials 2-10 (immediate visual memory), RULIT delayed recall scores, digit span (WAIS, sum of forwards, backwards, sequencing), symbol span (WMS), anti-saccades, flanker, and set-shifting (each from the EXAMINER battery).
Change in Functional Performance | After three months of training
  Between-group magnitude of change in sum time of all tasks in the Timed Instrumental Activities of Daily Living (TIADL). Higher scores indicate greater impairment in functional performance.

SECONDARY OUTCOMES:
Change in Mental Health-Related Quality of Life | After three months of training and 3 months after training completion
  Between-group magnitude of change in the Mental Component Score (MCS) as measured by the SF-12v2 Health Survey. The component score is a normed-based score with a mean of 50. Scores less than 50 indicate worse mental health than the mean.
Change in Physical Health-Related Quality of Life | After three months of training and 3 months after training completion
  Between-group magnitude of change in the Physical Component Score (PCS) as measured by the SF-12v2 Health Survey. The component score is a normed-based score with a mean of 50. Scores less than 50 indicate worse physical health than the mean.
Change in Depressive Symptoms | After three months of training and 3 months after training completion
  Between-group magnitude of change in sum score using the self-report measure, Beck Depression Inventory (BDI-II). The scoring range is 0-63. Higher scores indicate more severe depressive symptoms.
Change in PTSD Symptoms | After three months of training and 3 months after training completion
  Between-group magnitude of change in sum score using the self-report measure, PTSD Checklist - Civilian Version (PCL-C). The scoring range is 17-85. Higher scores indicate more severe PTSD symptoms.
Change in Executive Function Symptoms | After three months of training and 3 months after training completion
  Between-group magnitude of change in After total T-score using the self-report measure, Frontal Systems Behavior Scale (FrSBe). Raw scores are converted to age- and education-corrected T-scores. The mean T-score is 50, scores greater than 65 are considered clinically significant.
Change in Cognitive Symptoms | After three months of training and 3 months after training completion
  Between-group magnitude of change in sum score using the self-report measure, Cognitive Failures Questionnaire (CFQ). The scoring range is 0-100. Higher scores indicate more severe cognitive symptoms.
Change in Neurobehavioral Symptoms | After three months of training and 3 months after training completion
  Between-group magnitude of change in sum score using the self-report measure, Neurobehavioral Symptoms Index (NSI). The scoring range is 0-88. Higher scores indicate more severe neurobehavioral symptoms.
Change in TBI Functional Status | After three months of training and 3 months after training completion
  Between-group magnitude of change in overall T-score using the self-report measure, Mayo-Portland Adaptability Inventory (MPAI-4). The overall T-score range is -38 to 106. Higher scores indicate more severe TBI functional status.
Change in Immediate Verbal Memory | After three months of training and 3 months after training completion
  Between-group magnitude of change in sum of Trials 1-5 of the Rey Auditory Verbal Learning Test (RAVLT). The scoring range is 0-75. Lower scores indicate greater impairment in immediate verbal memory.
Change in Delayed Verbal Memory | After three months of training and 3 months after training completion
  Between-group magnitude of change in total score of delayed verbal recall on the Rey Auditory Verbal Learning Test (RAVLT). The scoring range is 0-15. Lower scores indicate greater impairment in delayed verbal memory.
Change in Immediate Visual Memory | After three months of training and 3 months after training completion
  Between-group magnitude of change in sum of Trials 2-10 of the Ruff Light Trails Test (RULIT). The scoring range is 0-135. Lower scores indicate greater impairment in immediate visual memory.
Change in Delayed Visual Memory | After three months of training and 3 months after training completion
  Between-group magnitude of change in total score of delayed visual recall on the Ruff Light Trails Test (RULIT). The scoring range is 0-15. Lower scores indicate greater impairment in delayed visual memory.
Change in Short-Term Verbal Memory Span | After three months of training and 3 months after training completion
  Between-group magnitude of change in sum of forwards, backwards, and sequencing tasks of the Wechsler Adult Intelligence Scale (WAIS) 4th Edition - Digit Span. The scoring range is 0-48. Lower scores indicate greater impairment in short-term verbal memory.
Change in Short-Term Visual Memory Span | After three months of training and 3 months after training completion
  Between-group magnitude of change in total score of the Wechsler Memory Scale (WMS) 4th Edition - Symbol Span. The scoring range is 0-50. Lower scores indicate greater impairment in short-term visual memory.
Change in Inhibition of Reflexive Saccade | After three months of training and 3 months after training completion
  Between-group magnitude of change in total score of the Anti-Saccade task of the Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER). The scoring range is 0-40. Lower scores indicate greater impairment in reflexive saccade inhibition.
Change in Response Inhibition | After three months of training and 3 months after training completion
  Between-group magnitude of change in total score of the Flanker task of the Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER). The scoring range is 0-10. Lower scores indicate greater impairment in response inhibition.
Change in Cognitive Flexibility | After three months of training and 3 months after training completion
  Between-group magnitude of change in total score of the Set-Shifting task of the Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER). The scoring range is 0-10. Lower scores indicate greater impairment in mental flexibility.
Change in Functional Performance | 3 months after training completion
  Between-group magnitude of change in sum score of all tasks in the Timed Instrumental Activities of Daily Living (TIADL). Higher scores indicate greater impairment in functional performance.

CONTACTS AND LOCATIONS:
Overall Officials: Henry W Mahncke, PhD, Principal Investigator — Posit Science Corporation; Cate N Stasio, BA, Study Director — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States

REFERENCES:
- [Background] Consensus conference. Rehabilitation of persons with traumatic brain injury. NIH Consensus Development Panel on Rehabilitation of Persons With Traumatic Brain Injury. JAMA. 1999 Sep 8;282(10):974-83. PMID 10485684